CLINICAL TRIAL: NCT02095327
Title: Religion and Free Will Perceptions as Coping Mechanisms in Caregivers of Individuals With Dementia
Brief Title: Families Affected by Dementia: A Survey of Caregivers
Acronym: FAD
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Amy Weisman, Associate Professor, University of Miami
Other Study IDs: 20130429
Record Dates: First submitted 2014-03-18; First posted 2014-03-24 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of our study is to better understand how caregivers of individuals with dementia cope with their family member's illness. If you are eligible for the study and would like to participate, we will schedule a one-time phone interview, which will last approximately 2 hours for which you will be compensated for your time.

DETAILED DESCRIPTION:
Eventually, results of this study will be used to develop treatments that will hopefully help caregivers cope more effectively with managing dementia in a loved one.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver of individual with dementia
* Relative who is 60 years or older with dementia
* Live-in, unpaid caregiver
* Have a working telephone number

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample of caregivers for individuals with dementia
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Depression | 3 months
  Measured continuously using the Depression, Anxiety and Stress Scale on a scale of 1 - 56.

SECONDARY OUTCOMES:
Anxiety | 3 months
  Measured continuously on the Depression, Anxiety, and Stress Scale on a scale of 1 - 56.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Weisman de Mamani, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

REFERENCES:
- See also: Visit our website for more information — https://plus.google.com/u/0/109687744987641360264/about